CLINICAL TRIAL: NCT03172455
Title: Early Access Program Using Alpha 1 Antitrypsin Infusion for Patients With Steroid Refractory Acute GvHD After Hematopoietic Stem Cell Transplantation (HSCT)
Status: No longer available | Type: Expanded Access
Sponsor: Impatients N.V. trading as myTomorrows (Industry)
Collaborators: Kamada, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-AATGLAKAM-EU
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Acute-graft-versus-host Disease; Steroid Refractory Acute Graft Versus Host Disease; Graft-versus-host-disease; Graft Vs Host Disease; Alpha 1-Antitrypsin Deficiency; Alpha-1 Proteinase Inhibitor; Alpha-1 Protease Inhibitor Deficiency; Acute Graft-Versus-Host Reaction Following Bone Marrow Transplant
MeSH Terms: conditions — Graft vs Host Disease; alpha 1-Antitrypsin Deficiency; alpha-1-Antitrypsin Deficiency, Autosomal Recessive | interventions — alpha 1-Antitrypsin

INTERVENTIONS:
Drug: Glassia — Application 90 mg/kg loading dose day 1, 30 mg/kg every other day (day 3 - day 15)
  Other Names: Alpha 1 antitrypsin

SUMMARY:
An Early Access Program for patients with steroid refractory acute GvHD after hematopoietic stem cell transplantation.

This Program is available for female and male who are recipients of allogenic HSCT and who have been newly diagnosed with acute GvHD.

DETAILED DESCRIPTION:
GLASSIA (human alpha-1 proteinase inhibitor (A1PI), also known as human alpha-1 antitrypsin, Kamada-AAT or Kamada-API) is a, liquid, ready-to-use preparation of human A1PI. Alpha-1 proteinase inhibitor belongs to the family of serine proteinase inhibitors and is primarily produced in the liver and secreted into the circulation. In addition to its anti-proteinase activity, A1PI showed to have anti-inflammatory, anti-apoptotic and immunomodulatory properties (1-4).

GLASSIA is an injection solution prepared from human plasma collected from healthy volunteer blood donors in accordance with Food and Drug Administration (FDA) and European Medicines Agency (EMA) regulations. GLASSIA was approved in the United States (US) in July 2010 and is indicated for chronic augmentation and maintenance therapy in adults with clinically evident emphysema due to severe hereditary deficiency of Alpha1-PI (alpha1-antitrypsin deficiency).

ELIGIBILITY:
Inclusion Criteria:

* This program is available for patients who suffer from steroid refractory acute GvHD after HSCT, or for whom, in the opinion of their treating physician, other treatment options or clinical trials in this indication are unsuitable.
* The disease indication for which the participant required HSCT must be in remission
* Acute graft-versus-host disease (aGvHD), including lower GI involvement (modified
* International Bone Marrow Transplant Registry (IBMTR) Severity Stage 1 to 4 [>500 mL diarrhea/day]), with or without other organ system involvement.
* For women of childbearing potential, had a negative serum or urine pregnancy test within 14 days prior to enrolment.

Exclusion Criteria:

* Participant with manifestations of chronic GvHD
* Participant with acute/chronic GvHD overlap syndrome
* Participant whose GvHD developed after donor lymphocyte infusion
* Participant with severe sepsis involving at least 1 organ failure
* Participant who is seropositive or positive in the nucleic acid test for human immunodeficiency virus (HIV)
* Participant with active hepatitis B or C
* If female, participant is pregnant or lactating at the time of enrollment, or has plans to become pregnant during the program

Sex: All
Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Background] Breit SN, Wakefield D, Robinson JP, Luckhurst E, Clark P, Penny R. The role of alpha 1-antitrypsin deficiency in the pathogenesis of immune disorders. Clin Immunol Immunopathol. 1985 Jun;35(3):363-80. doi: 10.1016/0090-1229(85)90097-2. PMID 3886224
- [Background] Toldo S, Seropian IM, Mezzaroma E, Van Tassell BW, Salloum FN, Lewis EC, Voelkel N, Dinarello CA, Abbate A. Alpha-1 antitrypsin inhibits caspase-1 and protects from acute myocardial ischemia-reperfusion injury. J Mol Cell Cardiol. 2011 Aug;51(2):244-51. doi: 10.1016/j.yjmcc.2011.05.003. Epub 2011 May 12. PMID 21600901
- [Background] Lewis EC, Mizrahi M, Toledano M, Defelice N, Wright JL, Churg A, Shapiro L, Dinarello CA. alpha1-Antitrypsin monotherapy induces immune tolerance during islet allograft transplantation in mice. Proc Natl Acad Sci U S A. 2008 Oct 21;105(42):16236-41. doi: 10.1073/pnas.0807627105. Epub 2008 Oct 13. PMID 18852465
- [Background] Churg A, Dai J, Zay K, Karsan A, Hendricks R, Yee C, Martin R, MacKenzie R, Xie C, Zhang L, Shapiro S, Wright JL. Alpha-1-antitrypsin and a broad spectrum metalloprotease inhibitor, RS113456, have similar acute anti-inflammatory effects. Lab Invest. 2001 Aug;81(8):1119-31. doi: 10.1038/labinvest.3780324. PMID 11502863